CLINICAL TRIAL: NCT05374187
Title: Efficacy of External Trigeminal Nerve Stimulation for Treatment of ADHD
Brief Title: Efficacy of Trigeminal Nerve Stimulation for ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James McGough, Professor of Clinical Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIHM R01 MH126041-01A1; 1R01MH126041-01A1 (NIH)
Record Dates: First submitted 2022-05-09; First posted 2022-05-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Attention-Deficit Hyperactivity Disorder
Keywords: ADHD; Neuromodulation; Trigeminal Nerve Stimulation; Cognition; EEG
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, sham-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active eTNS (Experimental): Following screening and determination of eligibility , participants at baseline are randomized to receive 4 weeks nightly treatment with active eTNS. Positive responders will be invited to participate in a 12-month open-label continuation phase.
  Interventions: Device: Active eTNS
- Sham eTNS (Sham Comparator): Following screening and determination of eligibility, participants at baseline are randomize to receive 4 weeks nightly treatment with sham eTNS. At conclusion of the double-blind phase, participants randomized to sham will be provided an opportunity to receive an additional 4 weeks nightly treatment with active eTNS. Positive responders to active eTNS will be invited to participate in a 12-month open-label continuation phase.
  Interventions: Device: Active eTNS; Device: Sham eTNS

INTERVENTIONS:
Device: Active eTNS — Participants will receive active trigeminal nerve stimulation (eTNS) administered by the Monarch eTNS system nightly during sleep for 4 weeks. Participants deemed to be positive responders to blinded active treatment will be invited to continue open nightly eTNS in a 12 month extension period.
  Other Names: Trigeminal Nerve Stimulation; Monarch eTNS SystemTM (NeuroSigma, Inc., Los Angeles, CA
Device: Sham eTNS — Participants will receive sham trigeminal nerve stimulation (eTNS) administered by the Monarch eTNS system nightly during sleep for 4 weeks. At conclusion of the blinded trial, participants randomized to the sham group will be offered 4 weeks of open active eTNS treatment. Participants deemed to be positive responders to open active treatment will be invited to continue open nightly eTNS in a 12 month extension period.
  Arms: Sham eTNS

SUMMARY:
This study is a large multisite randomized clinical trial to asses the efficacy of external trigeminal nerve stimulation (TNS), a novel, minimal risk, non-invasive neuromodulation treatment, for ADHD in children ages 7-12 years old (N=180).

Study hypotheses address potential differences in ADHD symptoms over 4 weeks treatment with active vs. sham TNS in an expanded multi-site investigation; whether resting state fronto-parietal connectivity mediates TNS impact on ADHD symptoms; if changes in fronto-parietal activation, as measured by electroencephalography (EEG), predict TNS-related treatment outcomes; and whether a baseline cognitive profile similarly predicts response to TNS therapy.

DETAILED DESCRIPTION:
Trigeminal Nerve Stimulation (TNS), an FDA-approved, non-invasive minimal risk intervention approved for treatment of Attention-Deficit/Hyperactivity Disorder (ADHD), administers a low amount of electrical stimulus to the forehead during sleep and is shown to increase activity in brain regions associated with attention and impulse control.

The current study seeks to replicate previous efficacy and safety findings of TNS in a larger, multisite group of ADHD-diagnosed youth, ages 7-12. The study will be conducted at UCLA and Seattle Children's Hospital.

The study comprises 3 phases, with subsequent 12-month follow-up for participants who demonstrate positive response to active therapy. We will screen up to 280 participants to yield an overall study N=225 completers meeting Diagnostic and Statistical Manual-5 (DSM-5) ADHD criteria across the two sites.

Phase 1 is a 4-week double-blind, controlled trial of active vs. sham TNS. Once inclusion/exclusion criteria are assessed, eligible participants have an initial baseline assessment comprised of behavioral ratings, cognitive assessments, and electroencephalography (EEG), and are subsequently randomized 2:1 to active vs. sham treatment. Participants will begin use of TNS as directed each night during sleep for 4 weeks. Participants, families, and most of the study team will remain blind to treatment assignment. Weekly behavioral rating will be obtained from parents, teacher, and clinical investigators. EEG, along with other cognitive measures, will be repeated at week 4.

In Phase 2, participants initially randomized to sham will receive active TNS for an additional 4 weeks, with continued weekly assessments. Phase 3 entails brief naturalistic follow-ups via phone or Zoom at months 3 and 6 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. male and female children ages 7 to 12 years with DSM-5 ADHD, any current presentation, as determined by diagnostic interview, Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS), and clinical interview;
2. total score >= 24 on baseline ADHD-RS;
3. CGI-S score at baseline >= 4;
4. no current medication with CNS effects (Participants previously on psychostimulant medication will be required to be not optimally treated and off medication for one week or 5 half-lives for all other medications); stable use of supplements will be permitted;
5. parents able and willing to monitor proper use of the stimulation device and complete all required rating scales;
6. estimated Full Scale IQ >= 80 based on WASI subtests;
7. parent and participant able to complete rating scales and other measures in English;
8. able to cooperate during EEG

Exclusion Criteria:

1. impaired functioning to a degree that requires immediate initiation of ADHD medication in the opinion of the parents and/or investigator;
2. current diagnosis of autism spectrum disorder or major depression;
3. history of lifetime psychosis, mania, or seizure disorder;
4. baseline suicidality;
5. history of seizure disorder or head injury with loss of consciousness

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD Rating Scale-5 (ADHD-RS-5) | Baseline, weeks 1, 2, 3, 4, 5, 6, 7, 8, 16, 20
  A dimensional rating of ADHD symptoms, with scores ranging from 0-54, and higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | Baseline, weeks 4, 8, 16, 20
  Categorical measure indicating overall degree of clinical severity among patients with similar diagnoses. Minimum score = 1 (Normal); Maximum score = 7 (Among the most extremely ill patients).
Clinical Global Impression - Improvement (CGI-I) | Weeks 1, 2, 3, 4, 5, 6, 7, 8, 16, 20
  Categorical measure indicating degree improved or not improved compared with baseline for each treatment group. Minimum score = 1 (very much improved); Maximum score = 7 (very much worse). Results reflect number of participants stratified as "Improved" (CGI-I <=2) or "Not Improved" (CGI-I > 2).
Change in Strengths and Weakness of Attention-Deficit/Hyperactivity (SWAN) Rating Scale | Baseline, weeks 1, 2, 3, 4, 5, 6, 7, 8, 16, 20
  A dimensional measure of ADHD symptoms measured on a 7-point scale, with scores ranging from -54 to +54, and lower scores indicating worse symptoms.
Change in Conners Short Form - Parent | Baseline, weeks 4, 8
  Parent completed dimensional measure of ADHD symptoms, with score range from 0-135, and higher scores indicating more severe symptoms.
Change in Conners Short Form - Teacher | Baseline, weeks 4, 8
  Teacher completed dimensional measure of ADHD symptoms, with score range from 0-123, and higher scores indicating more severe symptoms.
Change in Height | Baseline, weeks 4, 8
  A dimensional measure assessed in centimeters (cm).
Change in Weight | Baseline, weeks 4, 8
  A dimensional measure assessed in kilograms (kg).
Change in Weiss Functional Impairment Rating Scale | Baseline, weeks 4, 8
  A dimensional rating scale designed to evaluate the extent to which an individual's ability to function is impaired by emotional or behavioral problems, with scores ranging from 0 to 150, and higher scores signifying worse impairment.
Change in Child Depression Inventory | Baseline, weeks 4, 8
  A child completed dimensional rating of depressive symptoms, with scores ranging from 0 to 54, with higher scores indicating greater severity of depressive symptoms.

OTHER OUTCOMES:
Change in Electroencephalography (EEG) | Baseline, weeks 4, 8, 16
  A laboratory of cortical activity.
Change in Attention Network Task - Go/NoGo | Baseline, weeks 4, 8
  A computerized laboratory measure of response inhibition.
Change in Behavior Rating Inventory of Executive Functioning (BRIEF) | Baseline, weeks 1, 2, 3, 4, 5, 6, 7, 8, 16, 20
  A parent completed rating of child executive function. Comprises 5 sub scales that measure various measures of behavior and cognition. Raw scores on each measure are converted to T scores ran ging from 28 to 103, with higher scores indicating greater difficulties.
Change in Children's Sleep Habits Questionnaire (CSHQ) | Baseline, weeks 1, 2, 3, 4, 5, 6, 7, 8, 16, 20
  A parent completed 33-item scale to assess sleep related problems. Total scores range from 33 to 99 divided among 8 subscales, with higher scores indicating more severe difficulties.
Change in Happy CaFE | Baseline, weeks 4, 8
  A computerized task of emotional reactivity administered in conjunction with EEG

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K. Loo, Ph.D., Principal Investigator — University of California, Los Angeles; James J. McGough, M.D., Principal Investigator — University of California, Los Angeles; Mark A. Stein, Ph.D., Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The study will be registered on clinicaltrials.gov and all data will be uploaded to the National Database for Clinical Trials (NDCT) related to Mental Illness. Final de-identified data will be uploaded to NDCT databases by the PIs and trained research personnel at the completion of the study. All research data will be redacted to prevent the disclosure of personal identifiers.
  All individual participant data collected during the trial will be shared, following de-identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years after study publication.
Access Criteria: External investigators will be able to apply for access via an online query system by submitting their affiliations and details of their proposed research.

REFERENCES:
- [Background] McGough JJ, Loo SK, Sturm A, Cowen J, Leuchter AF, Cook IA. An eight-week, open-trial, pilot feasibility study of trigeminal nerve stimulation in youth with attention-deficit/hyperactivity disorder. Brain Stimul. 2015 Mar-Apr;8(2):299-304. doi: 10.1016/j.brs.2014.11.013. Epub 2014 Nov 28. PMID 25533244
- [Background] McGough JJ, Sturm A, Cowen J, Tung K, Salgari GC, Leuchter AF, Cook IA, Sugar CA, Loo SK. Double-Blind, Sham-Controlled, Pilot Study of Trigeminal Nerve Stimulation for Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2019 Apr;58(4):403-411.e3. doi: 10.1016/j.jaac.2018.11.013. Epub 2019 Jan 28. PMID 30768393
- [Background] McGough JJ, Loo SK, Cook IA. Reply to "Transcutaneous electric currents to target the peripheral and central nervous system in children with attention deficit hyperactivity disorder". Clin Neurophysiol. 2019 Oct;130(10):2008-2009. doi: 10.1016/j.clinph.2019.07.012. Epub 2019 Jul 23. No abstract available. PMID 31377119
- [Background] Loo SK, Salgari GC, Ellis A, Cowen J, Dillon A, McGough JJ. Trigeminal Nerve Stimulation for Attention-Deficit/Hyperactivity Disorder: Cognitive and Electroencephalographic Predictors of Treatment Response. J Am Acad Child Adolesc Psychiatry. 2021 Jul;60(7):856-864.e1. doi: 10.1016/j.jaac.2020.09.021. Epub 2020 Oct 15. PMID 33068751